CLINICAL TRIAL: NCT04095221
Title: A Phase I/II Dose Escalation/Dose Expansion Study of Prexasertib in Combination With Irinotecan in Patients With Relapsed or RefractoryDesmoplastic Small Round Cell Tumor and Rhabdomyosarcoma
Brief Title: A Study of the Drugs Prexasertib, Irinotecan, and Temozolomide in People With Desmoplastic Small Round Cell Tumor and Rhabdomyosarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-120
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Desmoplastic Small Round Cell Tumor; Rhabdomyosarcoma
Keywords: Prexasertib; Irinotecan; Temozolomide; 19-120
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor; Rhabdomyosarcoma | interventions — prexasertib; Irinotecan

STUDY DESIGN:
Intervention Model Description: This is a single institution study to determine the recommended phase 2 dose of prexasertib when given in combination with irinotecan and temozolomide. Patients with relapsed or refractory desmoplastic small round cell tumor or rhabdomyosarcoma of any subtype will receive prexasertib using the 3+3 dose-escalation schema.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prexasertib and Irinotecan (Experimental): Patients will have extent of disease scans following every 2 cycles (every 6 weeks on dose levels 0-3, and every 8 weeks on dose level -1 (if required). Patients will be allowed to continue therapy as long as they do not experience dose-limiting toxicities or progression of disease.
  Interventions: Drug: Prexasertib; Drug: Irinotecan

INTERVENTIONS:
Drug: Prexasertib — DOSE LEVELS FOR PATIENTS > 21 YEARS OF AGE, Dose Level -1, prexasertib 105 mg/ m2 once every 14 days in 28 day cycles Dose Level 0, 60 mg/m2 prexasertib once every 21 days Dose Level 1, (STARTING) 80 mg/m2 prexasertib once every 21 days Dose Level 2, 105 mg/m2 prexasertib once every 21 days Dose Level 3, 105 mg/m2 prexasertib once every 21 days
  DOSE LEVELS FOR PATIENTS ≤ 21 YEARS OF AGE Dose Level -1, prexasertib 150 mg/ m2 once every 14 days in 28 day cycles, Dose Level 0, 60 mg/m2 prexasertib once every 21 days, Dose Level 1, (STARTING) 80 mg/m2 prexasertib once every 21 days, Dose Level 2, 150 mg/m2 prexasertib once every 21 days, Dose Level 3, 150 mg/m2 prexasertib once every 21 days
Drug: Irinotecan — 15 mg/m2 IV daily x 10 days in 21 day cycles

SUMMARY:
The purpose of this study is to test whether the study drug prexasertib is a safe and effective treatment for people with DSRCT or RMS when given in combination with the standard drugs irinotecan and temozolomide. The study will test different doses of prexasertib in combination with irinotecan and temozolomide to find the highest dose of prexasertib that causes few or mild side effects in participants.

ELIGIBILITY:
Inclusion Criteria:

* Consent/Assent: all patients and/or their parents or legally authorized representatives must sign written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Age: patients must be ≥12 months of age at the time of study enrollment
* Diagnosis: patients must have histologically documented locally advanced or metastatic desmoplastic small round cell tumor or rhabdomyosarcoma (confirmed at MSK)
* Therapeutic options: patient's current disease state must be one which has failed standard therapy and for which there is no known curative therapy
* Disease Status: patients must have measurable disease based on RECIST 1.1
* Performance level: Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age
* Prior Therapy: patients may have had any number of prior therapies, but must have recovered from the acute toxic effects of all prior anti-cancer therapy (other than alopecia) as described below and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment

  °patients who have previously received irinotecan and/or temozolomide will be allowed
  * 21 days must have elapsed after the last dose of cytotoxic or myelosuppressive chemotherapy
  * 7 days must have elapsed after the last dose of anti-cancer agents not known to be myelosuppressive
  * 14 days must have elapsed after radiation therapy, and toxicity related to prior radiation therapy must be recovered to grade ≤ 1
  * 21 days must have elapsed after the last dose of antibody therapy, and toxicity related to prior antibody therapy must be recovered to grade ≤ 1
* Organ Function Requirements: Adequate bone marrow function defined as:

  * absolute neutrophil count (ANC) ≥ 1500/mm^3
  * platelet count ≥ 100,000/ mm^3
  * hemoglobin ≥ 8 g/dl
* Adequate renal function defined as:

  * Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min/1.73m2 OR
  * Serum creatinine based on age/gender derived from the Schwartz formula for estimating GFR53
* Adequate liver function defined as:

  * Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal for age
  * AST or ALT ≤ 5 x upper limit of normal for patients with liver metastases
  * Serum albumin ≥ 2.5 g/dl
* Adequate cardiac function defined as:

  * echocardiogram with left ventricular ejection fraction (LVEF) >45%
  * QTc < 470 ms on screening 12 lead electrocardiogram
* Pregnancy/Contraception

  * post-menarchal females must have a negative urine or serum pregnancy test at screening and ≤ 24 hours prior to study treatment
  * males or females of reproductive potential must be willing to use a barrier method of contraception throughout the course of the study and for 6 months after participation

Exclusion Criteria:

* Patients for whom the investigator deems that irinotecan and temozolomide are not appropriate are not eligible.
* Patients who have an uncontrolled infection are not eligible.
* Patients who are pregnant or breast feeding are not eligible.
* Patients who have a history of Torsades de Pointes, carry a diagnosis of congestive heart failure, or have a family history of prolonged QT syndrome are not eligible.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible.
* Patients with known hypersensitivity to irinotecan or its excipients are not eligible.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
recommended phase II does of Prexasertib | 1 year
  The RP2D is defined as the highest dose level associated with not more than 1 DLT out of 6 patients. A total of 5 dose levels are planned, including 2 back up levels. The DLT's will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The dose escalation will follow a 3+3 design.
response | 2 years
  will be evaluated in this study using the criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline, version 1.1 (Primary response criteria)54. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Slotkin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm